CLINICAL TRIAL: NCT02521610
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled, Ascending Dose Study to Investigate the Pharmacokinetics, Pharmacodynamic Effects, Safety and Tolerability of Repeated Dosing of RO5459072 in Healthy Subjects
Brief Title: A Multiple Ascending-Dose Study of RG7625 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BP29772
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Healthy volunteers will receive the placebo equivalent to RG7625 as oral capsules once or twice daily for 8 days. Each cohort will receive intradermal administration of 4 antigens (tetanus toxoid, tuberculin purified protein derivative [PPD], Candida albicans, and Trichophyton species) and a negative control at Screening and on Day 7 of treatment to assess for DTH.
  Interventions: Drug: Placebo
- RG7625 (Experimental): Participants will undergo a series of Screening visits prior to treatment and 7- to 14-day follow-up. Healthy volunteers will be enrolled in up to 4 cohorts and will receive RG7625 as oral capsules once or twice daily for 8 days. The first cohort is planned to receive 100 milligrams (mg) on Day 1, followed by 100 mg twice daily on Days 3 to 9. Subsequent dose and frequency decisions will be based upon observations in previous cohort(s). Each cohort will receive intradermal administration of 4 antigens (tetanus toxoid, tuberculin PPD, Candida albicans, and Trichophyton species) and a negative control at Screening and on Day 7 of treatment to assess for DTH.
  Interventions: Drug: RG7625

INTERVENTIONS:
Drug: Placebo — Participants will receive the placebo equivalent to RG7625 once or twice daily for 8 days. The first dose will be administered on Day 1 and the regimen will be continued during Days 3 to 9, with only a single dose given on Day 9.
  Arms: Placebo
Drug: RG7625 — Participants will receive RG7625 as oral capsules once or twice daily for 8 days. The first dose will be administered on Day 1 and the regimen will be continued during Days 3 to 9, with only a single dose given on Day 9.
  Arms: RG7625

SUMMARY:
This randomized, double-blind, placebo-controlled, ascending-dose, parallel-group study will evaluate the pharmacodynamic effects, pharmacokinetics, safety, and tolerability of one week of RG7625 dosing in healthy male and female volunteers. Each participant will receive a single dose of RG7625 or placebo followed by one week of dosing with the same treatment. Each participant will also receive intradermal administration of 4 recall antigens at Screening and on Day 7 of treatment to assess study drug effects on delayed-type hypersensitivity (DTH).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and females 18 to 60 years of age, inclusive
* Body mass index 18.0 to 30.0 kilograms per meter-squared (kg/m^2), inclusive

Exclusion Criteria:

* Any clinically relevant abnormalities, concomitant diseases or ongoing medical conditions, abnormal laboratory test results, or a history of any other clinically significant disorders
* Any major illness within the one month preceding the Screening visit, or any febrile illness within the two weeks preceding the Screening visit
* Any significant allergic reaction to drugs
* Immunocompromised or with reduced immune function and/or immunization within 30 days before the first study drug administration or planning vaccination during the study
* Women who are pregnant or lactating or of childbearing potential
* Clinically significant abnormal electrocardiogram (ECG) or other risk factors for QT prolongation
* Use of prescribed or over-the-counter medication
* Inability or unwillingness to comply with study requirements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in concentration of 10-kilodalton (kDa) cluster of differentiation (CD) 74 intermediate (p10) in B-cells | From Baseline (Day 1) to 24 hours after the Day 9 dose

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 9 weeks
Change in size of induration from DTH response | Up to 7 weeks
Area under the concentration-time curve (AUC) of RG7625 | Pre-dose at Baseline (Day 1) to 24 hours after the Day 9 dose
Maximum observed concentration (Cmax) of RG7625 | Pre-dose at Baseline (Day 1) to 24 hours after the Day 9 dose
Time to maximum observed concentration (Tmax) of RG7625 | Pre-dose at Baseline (Day 1) to 24 hours after the Day 9 dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands